CLINICAL TRIAL: NCT01234935
Title: A Multicenter, Open-Label, Randomized, Phase II Trial of Adjuvant Dasatinib Plus Gemcitabine Versus Single-Agent Gemcitabine in Patients With Resected Pancreatic Adenocarcinoma
Brief Title: Dasatinib and Gemcitabine Hydrochloride or Gemcitabine Hydrochloride Alone in Treating Patients With Pancreatic Cancer Previously Treated With Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Translational Oncology Research International (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRIO-TORI PA-01; NCI-2010-02190
Record Dates: First submitted 2010-11-01; First posted 2010-11-04 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Acinar Cell Adenocarcinoma of the Pancreas; Duct Cell Adenocarcinoma of the Pancreas; Recurrent Pancreatic Cancer; Stage IA Pancreatic Cancer; Stage IB Pancreatic Cancer; Stage IIA Pancreatic Cancer; Stage IIB Pancreatic Cancer; Stage III Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Dasatinib; Gemcitabine; Base Sequence; Immunohistochemistry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive gemcitabine hydrochloride IV on days 1, 8, and 15. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: gemcitabine hydrochloride; Other: laboratory biomarker analysis; Genetic: mutation analysis; Genetic: nucleic acid sequencing; Other: immunohistochemistry staining method
- Arm II (Experimental): Patients receive gemcitabine hydrochloride IV on days 1, 8, and 15 and oral dasatinib once daily on days 1-28. Treatment repeats every 28 days for 6 courses* in the absence of disease progression or unacceptable toxicity. NOTE: *Courses with dasatinib repeat every 28 days for 1 year in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: dasatinib; Drug: gemcitabine hydrochloride; Other: laboratory biomarker analysis; Genetic: mutation analysis; Genetic: nucleic acid sequencing; Other: immunohistochemistry staining method

INTERVENTIONS:
Drug: dasatinib — Given orally
  Other Names: BMS-354825; Sprycel
  Arms: Arm II
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; dFdCyd; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar; LY-188011
Other: laboratory biomarker analysis — Correlative studies
Genetic: mutation analysis — Correlative studies
Genetic: nucleic acid sequencing — Correlative studies
  Other Names: Gene Sequencing; Molecular Biology, Nucleic Acid Sequencing
Other: immunohistochemistry staining method — Correlative studies
  Other Names: immunohistochemistry

SUMMARY:
RATIONALE: Dasatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as gemcitabine hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. It is not yet known whether giving dasatinib together with gemcitabine hydrochloride is more effective than gemcitabine hydrochloride alone in treating pancreatic cancer. PURPOSE: This randomized phase II trial is studying how well giving dasatinib together with gemcitabine hydrochloride works compared to giving gemcitabine hydrochloride alone in treating patients with pancreatic cancer previously treated with surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. To compare disease-free survival at 18 months between dasatinib-gemcitabine combination therapy and single-agent gemcitabine. SECONDARY OBJECTIVES: I. To evaluate effects on disease-free survival of the dasatinib-gemcitabine combination therapy compared with gemcitabine alone for adjuvant treatment of resected pancreatic adenocarcinoma. II. To evaluate effects on overall survival of dasatinib-gemcitabine combination therapy compared with gemcitabine alone for adjuvant treatment of resected pancreatic adenocarcinoma. III. To evaluate tolerability and safety of the two arms. IV. To identify potential biological correlates associated with clinical benefit to dasatinib-gemcitabine combination therapy compared with gemcitabine alone. OUTLINE: Patients are randomized to 1 of 2 treatment arms. ARM I: Patients receive gemcitabine hydrochloride IV on days 1, 8, and 15. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity. ARM II: Patients receive gemcitabine hydrochloride IV on days 1, 8, and 15 and oral dasatinib once daily on days 1-28. Treatment repeats every 28 days for 6 courses* in the absence of disease progression or unacceptable toxicity. NOTE: * Courses with dasatinib repeat every 28 days for 1 year in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent before beginning any protocol specified procedures
* Histologically proven pancreatic adenocarcinoma
* Any T, any N, M0 disease that has had all gross disease resected (R0 or R1 resection)
* ECOG Performance status index 0 or 1
* Absolute Neutrophils >= 1.5 x 10^9/L
* Platelets >= 100 x 10^9/L
* Hemoglobin >= 10 g/dL
* Total bilirubin =< 2.0 x UNL; subjects with Gilbert's syndrome, confirmed by genotyping or invader UGTIA1 molecular assay before study entry must have total bilirubin < 3 x UNL
* ASAT (SGOT) and ALAT (SGPT) =< 2.5 x UNL
* Alkaline Phosphatase =< 5 x UNL
* Creatinine < 1.5 x UNL
* Serum Na, K+, Magnesium, Phosphate and Calcium >= LNL
* First study treatment must be given within 60 days after surgery and within 7 days after randomization
* Patients must be accessible for treatment and follow-up and compliant with study procedures
* Negative pregnancy test (urine or serum) within 7 days before first study treatment for all women of childbearing potential, whom also must implement adequate non-hormonal contraceptive measures during study treatment and for at least 3 months after the last dose of study therapy
* Ability to take oral medication (dasatinib must be swallowed whole)

Exclusion Criteria:

* Prior or concurrent systemic anticancer therapy (immunotherapy, hormonal therapy, biological therapy, or chemotherapy) for pancreatic cancer
* Prior or concurrent radiation therapy for pancreatic cancer
* Pregnant or lactating patients
* M1 pancreatic cancer
* Concurrent congestive heart failure, unstable angina pectoris, or M1 within the 6 months before first study treatment
* Uncontrolled hypertension or high-risk uncontrolled arrhythmias
* Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or torsades de pointes)
* Diagnosed or suspected congenital long QT syndrome
* Prolonged QTc interval on pre-entry electrocardiogram (> 450 msec)
* History of significant neurologic or psychiatric disorders including psychotic disorders, dementia or seizures that would prohibit the understanding and giving of informed consent
* Past or current history of neoplasm other than pancreatic adenocarcinoma, except for: curatively treated non-melanoma skin cancer; in situ carcinoma of the cervix; other cancer curatively treated and with no evidences of disease for at least 1 year
* Concurrent treatment with other experimental drugs or treatment with investigational drugs within 30 days of first study treatment
* Currently receiving drugs with known significant CYP 3A4 inhibitory effects (such as ketoconazole, itraconazole, troleandomycin, erythromycin, diltiazem, verapamil, ritonavir, indinavir)
* Concurrent administration with inducers of CYP 3A4 may result in a lower exposure to dasatinib and are therefore not allowed (e.g., phenytoin, carbamazepine, rifampicin, phenobarbital, pentobarbital, or St John's Wort)
* Known allergy reactions to dasatinib or gemcitabine or excipients used in the study
* History of significant bleeding disorders unrelated to cancer, including: diagnosed congenital bleeding disorders (e.g., Von Willebrand's disease); diagnosed acquired bleeding disorder within 1 year (e.g., acquired anti-factor VIII antibodies); ongoing or recent (=< 3 months) significant gastrointestinal bleeding
* Patients currently taking drugs that are generally accepted to have a risk of causing Torsades De Pointes including: quinidine, procainamide, disopyramide; amiodarone, sotalol, ibutilide, dofetilide; erythromycins, clarithromycin; chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide; cisapride, bepridil, droperidol, methadone, arsenic, chloroquine, domperidone, halofantrine, levomethadyl, pentamidine, sparfloxacin, lidoflazine
* Concurrent treatment with intravenous bisphosphonates; prior treatment should be stopped at least 2 weeks before first dose of study treatment
* Concurrent medical condition which may increase the risk of toxicity, including pleural or pericardial effusion or any grade
* Active uncontrolled infection requiring parenteral antimicrobials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-01-13 (Actual); Primary Completion 2017-11-27 (Actual); Study Completion 2017-11-27 (Actual)

PRIMARY OUTCOMES:
Disease-free survival | At 18 months

SECONDARY OUTCOMES:
Overall survival | follow-up every 3 months for 30 months from first treatment or until disease recurrence or withdrawal of consent
Disease-free survival | at 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard Finn, Principal Investigator — Translational Oncology Research International
Locations (17):
- United States (17):
  - Central Hematology Oncology Medical Group, Inc., Alhambra, California
  - TORI FULLERTON (St. Jude Heritage Healthcare Virginia K. Crosson Cancer Center), Fullerton, California
  - Pacific Shores Medical Group, Long Beach, California
  - UCLA medical center, Los Angeles, California
  - Translational Oncology Research International (TORI) Network, Los Angeles, California
  - TORI NORTHRIDGE (North Valley Hematology/Oncology Medical Group), Northridge, California
  - UCLA Pasadena, Pasadena, California
  - TORI Inland Valley (Wilshire Oncology Medical Group, Inc. ), Pomona, California
  - TORI REDONDO BEACH (Cancer Care Associates Medical Group, Inc.), Redondo Beach, California
  - TORI SANTA BARBARA I (Santa Barbara Hematology Oncology Medical Group, Inc.), Santa Barbara, California
  - TORI SANTA BARBARA II (SANSUM Clinic), Santa Barbara, California
  - TORI SANTA MARIA (Central Coast Medical Oncology Corporation), Santa Maria, California
  - UCLA Valencia, Valencia, California
  - Suburban Hematology-Oncology Associates, P.A., Lawrenceville, Georgia
  - Northwest Georgia Oncology Centers, P.C., Marietta, Georgia
  - Chevy Chase Healthcare Management, LLC, Chevy Chase, Maryland
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada